CLINICAL TRIAL: NCT05614973
Title: Efficacy and Safety of Percutaneous Liver Biopsy With Needle Tract Plugging on Outpatient Basis: a Randomized Study (COGEL Study; Coaxial With Gelatin)
Brief Title: Efficacy and Safety of Percutaneous Liver Biopsy With Needle Tract Plugging on Outpatient Basis
Acronym: COGEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2022-0211
Record Dates: First submitted 2022-11-01; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Image-guided Biopsy; Liver Biopsy

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be randomly allocated to either the conventional group or coaxial/plugging group for percutaneous liver biopsy. After the procedure, the rates of biopsy-related complications as well as diagnostic yield will be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Percutaneous liver biopsy is carried out through multiple punctures of liver capsule.
  Interventions: Procedure: Conventional method
- Coaxial/plugging (Experimental): Percutaneous liver biopsy is carried out through single puncture of liver capsule using coaxial needle and subsequent needle tract plugging.
  Interventions: Procedure: Coaxial method with needle-track plugging

INTERVENTIONS:
Procedure: Conventional method — The conventional method utilizes a 18G biopsy gun to acquire three or more tissue cores with the corresponding number of liver capsule punctures. Plugging of the biopsy needle track is not performed.
  Arms: Conventional
Procedure: Coaxial method with needle-track plugging — The coaxial method utilizes a 17G coaxial needle with 18G biopsy gun to acquire three or more tissue cores with a single liver capsule puncture. Biopsy needle track is plugged using a slurry of gelatin particles (EGgel S Plus 2000-4000 μm).
  Arms: Coaxial/plugging

SUMMARY:
A prospective, randomized, two-arm, single-center study to compare efficacy and safety of percutaneous ultrasound-guided liver biopsy of conventional method (multiple liver punctures) versus coaxial method followed by needle tract plugging.

DETAILED DESCRIPTION:
Adult patients who are referred for the ultrasound-guided percutaneous biopsy of focal liver lesion (larger than 1cm) to obtain three or more tissue cores are eligible for this study. Exclusion criteria are as follows: 1) unable to approach a target lesion under ultrasound-guidance; 2) severe coagulopathy; 3) unable to discontinue anticoagulant/antiplatelet medications for the duration proposed by 2019 Society of Interventional Radiology guidelines; 4) co-presence of amyloidosis, large amount of ascites, or acute hepatobiliary infections. All enrolled patients will be randomized into either the conventional group or coaxial/plugging group. The conventional group will undergo percutaneous liver biopsy for multiple tissue cores through multiple punctures of the liver capsule. The coaxial/plugging group will undergo percutaneous liver biopsy using a coaxial needle (single puncture of the liver capsule), which will be plugged by gelatin particles after obtaining multiple tissue cores. The biopsy will be performed on outpatient basis regardless of the randomized group, and the patients will be discharged after two hours of observation. The rate of biopsy-related complications including bleeding (minor and major) and diagnostic yield will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. All adult patients aged 19 years or older in this institution
2. Patients referred for imaging-guided percutaneous liver biopsy requiring three or more tissue cores
3. Patients who understand and consent to enrollment in this study
4. Target lesion diameter 1cm or larger, and the lesion is approachable under ultrasonography-guidance.

Exclusion Criteria:

1. Patients with severe psychologic disorder or mental retardation
2. Patients with poor cooperation
3. Severe coagulopathy
4. Hepatobiliary obstruction
5. Acute hepatobiliary infection
6. Large amount of ascites
7. Amyloidosis
8. Patients on antiplatelet/anticoagulant medication that cannot be discontinued for a specified period of time
9. Other patients whom the researchers deem ineligible

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety of percutaneous liver biopsy | During procedure
  Biopsy-related bleeding
  * Minor bleeding is defined as presence of linear flow signal along the needle tract on Doppler exam.
  * Major bleeding is defined as bleeding which requires transfusion or vascular embolization.
Safety of percutaneous liver biopsy | Day 1 after procedure
  Biopsy-related bleeding
  * Minor bleeding is defined as presence of linear flow signal along the needle tract on Doppler exam.
  * Major bleeding is defined as bleeding which requires transfusion or vascular embolization.
Safety of percutaneous liver biopsy | Day 7 after procedure
  Biopsy-related bleeding
  * Minor bleeding is defined as presence of linear flow signal along the needle tract on Doppler exam.
  * Major bleeding is defined as bleeding which requires transfusion or vascular embolization.

SECONDARY OUTCOMES:
Efficacy of percutaneous liver biopsy | 1 week
  Number of successfully acquired tissue cores; Diagnostic yield

CONTACTS AND LOCATIONS:
Overall Officials: Seung-seob Kim, Principal Investigator — Severance hospitalDepartment of Radiology, Severance Hospital, Yonsei University College of Medicine, Korea
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea